CLINICAL TRIAL: NCT07370974
Title: Effect of Clinical Hypnosis in Preoperative Anxiety Among Patients Undergoing an Abdominal Surgery : a Multicenter Randomized Controlled Trial.
Brief Title: Effect of Clinical Hypnosis in Preoperative Anxiety Among Patients Undergoing an Abdominal Surgery.
Acronym: Hypnoanxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HASSAN 1st university (Other)
Responsible Party: Principal Investigator, YOUSSEF EL-ALLAM, Principal investigator, HASSAN 1st university
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Hypnosis UHP
Record Dates: First submitted 2026-01-02; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Hypnosis; Preoperative Anxiety; Postoperative Pain; Abdominal Surgeries; Length of Stay
Keywords: RCT; Morocco; Hypnosis; preoperative anxiety
MeSH Terms: conditions — Pain, Postoperative | interventions — Hypnosis

STUDY DESIGN:
Masking Description: This study did not use any kind of masking or blinding,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fisrt arm: patients having a session of hypnosis prior to surgery (Experimental): Patients randomized to the intervention arm undergo a single 15-20 minute clinical hypnosis session preoperatively for anxiety reduction, achieving level 2 hypnotic trance (somnambulism)
  Interventions: Other: Clincal hypnosis
- Arm 2 : patients will be treated as usual with standard conditions (No Intervention): Patients in this group will receive standard usual care without any hypnotic intervention, only with routine psychological preparation.

INTERVENTIONS:
Other: Clincal hypnosis — Patients randomized to the intervention arm receive a single 15-20 minute individual clinical hypnosis session 30-60 minutes preoperatively. The standardized protocol includes:
  * Induction phase (3-5 min): Eye fixation, progressive relaxation breathing
  * Deepening phase (5 min): Level 2 somnambulistic trance achievement
  * Therapeutic suggestions (7-10 min): Anxiety reduction imagery, surgical calm visualization
  * Emergence phase (2-3 min): Safe awakening to alert consciousness
  Delivered by certified hypnotherapist using validated script for preoperative anxiety in abdominal surgery patients." Key Elements Required Timing: Preop holding area, 30-60 min before incision Provider: Trained clinician (specify certification) Dose: Single 15-20 min session Target: Level 2 hypnosis (somnambulism) Outcome link: EVA anxiety scale pre/post This matches your 3-center RCT design (~16 patients/center, stratified randomization) and distinguishes from control arm (standard psychological preparation
  Other Names: Hypnosis, hypnotism; Hypnosis session
  Arms: Fisrt arm: patients having a session of hypnosis prior to surgery

SUMMARY:
This Multicenter randomized controlled trial evaluates clinical hypnosis efficacy for reducing perioperative anxiety and postoperative pain in abdominal surgery patients across 3 Moroccan centers (n=48-68). Intervention arm receives 15-20 min level 2 hypnosis session preoperatively; control receives standard psychological preparation. Primary outcome: VAS-anxiety post-intervention. Secondary: postoperative EVA-pain, analgesic consumption, length of stay.

Study Design Prospective, multicenter, parallel-group RCT (1:1 allocation, stratified by center/sex). Inclusion: consenting ASA I-II adults for abdominal surgery. Primary endpoint powered for 10mm EVA reduction (80% power, α=0.05). Registration supports PhD thesis at ISSS/Université Hassan 1er Settat.

ELIGIBILITY:
* Inclusion Criteria:

  1. Consenting patients undergoing abdominal surgery
  2. ASA I-II physical status
  3. Able to understand and respond to instructions
  4. No major psychological disorders
* Exclusion Criteria:

  1. Non-consenting patients
  2. Prior experience with hypnosis
  3. History of mental illness
  4. Psychoactive substance consumption
  5. Cognitive disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Preoperative anxiety | 1 hour Before surgery
  Perioperative Anxiety (Primary Outcome) is measured using the Visual Analog Scale for Anxiety (EVA-Anxiété, 0-100 mm).
  Primary Outcome Measure: preoperative anxiety level
  Assessment Tool: 100-mm Visual Analog Scale (VAS-Anxiety):
  0 mm = No anxiety ("Je ne suis pas du tout anxieux") 100 mm = Worst possible anxiety ("Anxiété maximale imaginable") Timepoints: (post-intervention, ~10 min later). Expected hypnosis effect: ≥10 mm reduction vs. control.
  Protocol Specifications Patient marking: Single horizontal 100-mm line; mark position indicates intensity Scoring: Distance (mm) from "No anxiety" (0) to mark, precise to 1 mm

SECONDARY OUTCOMES:
Postoperative pain | 6 and 24 hours postoperatively
  Secondary Outcome Measure: Acute postoperative pain intensity at 6, and 24 hours post-surgery.
  Assessment Tool: 100-mm VAS-Pain Scale:
  0 mm = No pain ("Aucune douleur") 100 mm = Worst imaginable pain ("Douleur maximale imaginable") Timepoints: T+6h, T+24h. Expected hypnosis benefit: ≥10 mm reduction vs. control .
  Protocol Specifications Patient marking: Horizontal 100-mm line; precise mm measurement from 0 Analgesia standardization: Multimodal protocol identical across arms (paracetamol, NSAIDs, opioids rescue) Power: Secondary analysis leverages primary outcome sample (48-68 patients, 80% power for Δ=10 mm, σ=24 mm)
  ClinicalTrials.gov Entry: "Postoperative pain intensity measured by 100-mm Visual Analog Scale at rest in PACU at 1, 2, 6, and 24 hours post-surgery"
  This complements your prim
medication consumption | Perioperative
  Secondary Outcome Measure: Anesthia drugs consumption and postoperative consumption of analgesics (morphine equivalents, paracetamol, NSAIDs, opioids) from PACU arrival to discharge.
  Assessment Method:
  Total mg/doses per patient, Data collection: Medication administration records (MAR), nurse logs Expected hypnosis effect: ≥20-30% reduction vs. control arm. Protocol Specifications
  Standardized multimodal analgesia (identical both arms):
length of stay | Perioperative
  Secondary Outcome Measure: Time to hospital discharge (days) from surgery day (Day 0) to medical discharge order date.
  Assessment Method:
  Calendar days: Date of discharge hour date of surgery Expected hypnosis effect: ≥1 day reduction vs. control (typical LOS 3-5 days abdominal surgery).
  Protocol Specifications
  Standardized discharge criteria (identical both arms):
  Tolerates solid diet VAS-pain ≤30 mm at rest Mobilizes independently to bathroom Afebrile, normal vital signs Data collection: medical record discharge order timestamp

CONTACTS AND LOCATIONS:
Overall Officials: NAOUFAL HIMMOUCHE HIMMOUCHE, Professor, Study Director — Laboratory of health sciences and technlmogies, Higher Institute of Health sciences, Hassan Fisrt University, Settat Morocco; YASSINE HAFIANI, Professor, Study Director — Pedagogical Unit of Anesthesia and Intensive Care, Rabat Faculty of Medicine and Pharmacy, Mohammed V University, Rabat, Morocco
Locations (3):
- Morocco (3):
  - Kenitra, Rabat Sale Kenitra region, Morocco, Kenitra, Province
  - Settat, Casablanca settat region , Morocco, Settat, Province
  - Youssoufia, Marrakech-Safi Morocco, Youssoufia, Province

IPD SHARING:
Plan to Share IPD: No
Data sharing not planned. Individual patient data will not be shared due to:" Small sample size (n=60 across 3 centers) creates high re-identification risk in Morocco's healthcare context Patient consent forms obtained pre-NIH Policy 2.0 did not include data sharing provisions Doctoral thesis protocol approved by CERB Mohammed V Rabat without data sharing plan Local data protection regulations (Loi 28-13) limit identifiable health data transfer Resource constraints prevent data de-identification and controlled access infrastructure Summary results, statistical analysis plan, and blinded protocol available upon request to corresponding author post-publication.